CLINICAL TRIAL: NCT00729755
Title: Efficacy and Safety of Augmentation of Creatine for the Patients With Major Depressive Disorder
Brief Title: Creatine Augmentation Treatment in Major Depressive Disorder Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIC-08DE00101B
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Major Depressive Disorder
Keywords: Creatine; Augmentation; Major Depressive Disorder; Efficacy; Brain Energy Metabolism
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Creatine (Experimental): The subjects with major depressive disorder, treated with creatine in addition to escitalopram
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): The subjects with major depressive disorder, treated with placebo in addition to escitalopram
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — In addition to 10-20mg escitalopram, the subjects will be given total 3 gram of creatine (500mg/capsule) a day in first week and then, 5 gram a day in the rest of the weeks.
  Arms: Creatine
Dietary Supplement: Placebo — In addition to 10-20mg escitalopram, the subjects will be given total 6 capsules of placebo (equal quantities to those of creatine group) a day in first week and then, 10 capsules a day in the rest of the weeks.
  Arms: Placebo

SUMMARY:
Given 1) the established safety with short-term or long-term supplementation of Cr, 2) its potential usefulness in improving brain energy metabolism, 3) the reported abnormality in brain energy metabolism in MDD subjects, and 4) plausible association between depression and inflammatory mediators, we hypothesize that oral Cr augmentation will help reduce symptoms in MDD patients as well as normalize a deficit in brain energy metabolism and that improvement of MDD and brain energy metabolism will be correlated with inflammatory mediators changes.

In this study, we plan to conduct an randomized, double-blind, placebo-controlled augmentation study with creatine in addition to escitalopram. We will assess the efficacy and safety of the Cr augmentation and evaluate changes relevant to brain energy metabolism and inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 year-old male or female
* Major depressive disorder diagnosed by SCID-IV
* Hamilton depression rating scale score >= 16 at screening
* Written informed consent

Exclusion Criteria:

* Suicidal idea that needs hospitalization
* Any other axis I psychiatric disorder
* Neurologic disease (eg., epilepsy, infarct, multiple sclerosis, brain tumor)
* IQ below 80
* Inflammatory disease including autoimmune disease
* Taking anti-inflammatory medication
* Serious physical disease
* Substance abuse or dependence history in recent 6 months
* Pregnant or having plan to be pregnant

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating scale | baseline, 1st, 2nd, 4th, 8th week

SECONDARY OUTCOMES:
Clinical global impression scale | baseline, 1st, 2nd, 4th, 8th week
Side effects assessment: the interview and examination by the investigators | baseline, 1st, 2nd, 4th, 8th week
Serum inflammatory mediators (eg., IL-1, -2, PGE2, interferon gamma) level | baseline, 8th week
Serum creatinine level | baseline, 2nd, 8th week
Brain MRI | baseline, 8th week
Montgomery-Asberg depression scale | baseline, 1st, 2nd, 4th, 8th week

CONTACTS AND LOCATIONS:
Overall Officials: Perry F Renshaw, MD, PhD, Study Chair — University of Utah; In Kyoon Lyoo, MD, PhD, MMS, Study Director — Ewha Womans University
Locations (4):
- South Korea (4):
  - Holy Family Hospital, Bucheon-si, Gyeonggi-do
  - Seoul St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - St. Paul's Hospital, Seoul

REFERENCES:
- [Derived] Yoon S, Kim JE, Hwang J, Kim TS, Kang HJ, Namgung E, Ban S, Oh S, Yang J, Renshaw PF, Lyoo IK. Effects of Creatine Monohydrate Augmentation on Brain Metabolic and Network Outcome Measures in Women With Major Depressive Disorder. Biol Psychiatry. 2016 Sep 15;80(6):439-447. doi: 10.1016/j.biopsych.2015.11.027. Epub 2015 Dec 15. PMID 26822799
- [Derived] Lyoo IK, Yoon S, Kim TS, Hwang J, Kim JE, Won W, Bae S, Renshaw PF. A randomized, double-blind placebo-controlled trial of oral creatine monohydrate augmentation for enhanced response to a selective serotonin reuptake inhibitor in women with major depressive disorder. Am J Psychiatry. 2012 Sep;169(9):937-945. doi: 10.1176/appi.ajp.2012.12010009. PMID 22864465